CLINICAL TRIAL: NCT03923114
Title: iPAVE - Imaging Pituitary ActiVation by Exendin
Brief Title: Imaging Pituitary ActiVation by Exendin
Acronym: iPAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL67316.091.18
Record Dates: First submitted 2019-04-11; First posted 2019-04-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: exendin; GLP-1 receptor agonist; HPA-axis; Imaging
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group with treatment response (Other): PET/CT imaging of patients with response to GLP-1 receptor agonist treatment
  Interventions: Radiation: Ga-68-NODAGA-exendin-4 PET/CT
- Patient group without treatment response (Other): PET/CT imaging of patients with no response to GLP-1 receptor agonist treatment
  Interventions: Radiation: Ga-68-NODAGA-exendin-4 PET/CT

INTERVENTIONS:
Radiation: Ga-68-NODAGA-exendin-4 PET/CT — PET/CT imaging after injection with Ga-68-NODAGA-exendin-4

SUMMARY:
The main goal is the comparison of pituitary uptake of Ga-68-NODAGA-exendin-4 in patients with and without adequate response (based on HbA1c or weight loss) to GLP-1R agonist treatment.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes (T2D) is increasing and a better understanding of the mechanisms of T2D becomes increasingly important. The glucagon-like peptide 1 receptor agonists (GLP-1RA), such as exendin, can be used as potent antidiabetic drugs for treatment of T2D. Not all patients with T2D respond to treatment with GLP-1RA and some even respond with contradictory effects, but the underlying mechanism for this observation remains unclear. Interestingly, uptake of an exendin-based radiotracer was observed in the pituitary gland in diabetes patients. In this study, the effect of GLP-1RA on the HPA axis will be further studied for an improved understanding of the mechanisms and contradictory treatment responses.

Patient data will be obtained and will consist of metabolic characterization (laboratory parameters and oral glucose tolerance test), an ACTH assay and determination of cortisol excretion. In addition, Ga-68-NODAGA-exendin-4 PET/CT imaging will be performed in 10 patients with treatment response (decrease in HbA1c or weight loss) and 10 patients without response after GLP-1RA therapy. In 5 patients with high radiotracer uptake, an additional brain MRI scan will be performed for improved anatomical referencing.

ELIGIBILITY:
Inclusion Criteria:

Patients with treatment response:

* Age ≥18 years
* Subject is diagnosed with type 2 diabetes
* Subject showed response to GLP-1RA treatment
* Ability to sign informed consent

Patients without treatment response:

* Age ≥18 years
* Subject is diagnosed with type 2 diabetes
* Subject showed no response to GLP-1RA treatment
* Ability to sign informed consent

Exclusion Criteria:

* Liver disease
* Renal disease
* Pregnancy or the wish to become pregnant within 6 months after the study
* Breastfeeding
* Age <18 years
* Pituitary disorder
* Inability to sign informed consent
* Exclusion criteria for MR:

  * Fragments, clips or devices in brain, eyes, spinal canal
  * Implantable defibrillator or pacemaker (wires)
  * Mandibular magnetic implants
  * Neurostimulator, bladder stimulator, non-removable insulin pump
  * Metal tissue-expander in chest
  * Cochlear implant
  * Ossicular replacement prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Pituitary uptake of Ga-68-NODAGA-exendin | 1.5 year
  Comparison of the pituitary uptake (Bq) of Ga-68-NODAGA-exendin-4 obtained by quantitative analysis

SECONDARY OUTCOMES:
Metabolic status (OGTT) | 1.5 year
  Assessment of the metabolic status by performing an OGTT (mmol/l)
Metabolic status (ACTH) | 1.5 year
  Assessment of the metabolic status by performing an ACTH assay (mol/l)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No